CLINICAL TRIAL: NCT02891824
Title: A Randomized, Double-blinded, Phase III Study of Atezolizumab Versus Placebo in Patients With Late Relapse of Epithelial Ovarian, Fallopian Tube, or Peritoneal Cancer Treated by Platinum-based Chemotherapy and Bevacizumab
Brief Title: ATALANTE: Atezolizumab vs Placebo Phase III Study in Late Relapse Ovarian Cancer Treated With Chemotherapy+Bevacizumab
Acronym: ATALANTE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ARCAGY/ GINECO GROUP (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GINECO-OV236b
Record Dates: First submitted 2016-05-25; First posted 2016-09-08 (Estimated); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Ovarian Cancer
Keywords: PD-L1; Atezolizumab; Randomized, double blinded; first or second late relapse; progressive non-mucinous epithelial ovarian cancer, primary peritoneal adenocarcinoma and / or fallopian-tube adenocarcinoma; progression-free survival
MeSH Terms: conditions — Ovarian Neoplasms | interventions — atezolizumab; Bevacizumab; Platinum Compounds

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Placebo + Avastin + platinum-based chemotherapy (Placebo Comparator): The placebo arm:
  Placebo 1200 mg x 6 cycles q3wk or 800mg x 6 cycles q4wk during treatment with chemotherapy and Avastin, followed by placebo 1200mg q3wk until progression
  Interventions: Drug: placebo + avastin + platinum-based chemotherapy
- Arm B: Atezolizumab + Avastin+ platinum-based chemotherapy (Experimental): The atezolizumab arm:
  Atezolizumab 1200 mg x 6 cycles q3wk or 800mg x 6 cycles q4wk during treatment with chemotherapy and Avastin, followed by atezolizumab 1200mg q3wk until progression
  .
  Interventions: Drug: atezolizumab + avastin + platinum-based chemotherapy

INTERVENTIONS:
Drug: atezolizumab + avastin + platinum-based chemotherapy — * atezolizumab will be administrated by intraveinous route at dose of 1200 mg or 800 mg during the induction period and will be continued in maintenance period at a dose of 1200mg until progression
  * avastin will be administrated by intraveinous route at dose of 15mg/kg or 10 mg/kg during the induction period and will be continued in maintenance period of at a dose of 15mg/kg until progression
  * platinum-based chemotherapy (Carboplatin combined with gemcitabine or paclitaxel or pegylated liposomal doxorubicin) will be administrated by intraveinous route at different doses during the induction period x 6 cycles
  Other Names: Tecentriq
  Arms: Arm B: Atezolizumab + Avastin+ platinum-based chemotherapy
Drug: placebo + avastin + platinum-based chemotherapy — * placebo will be administrated by intraveinous route at dose of 1200 mg or 800 mg during the induction period and will be continued in maintenance period at a dose of 1200mg until progression
  * avastin will be administrated by intraveinous route at dose of 15mg/kg or 10 mg/kg during the induction period and will be continued in maintenance period of at a dose of 15mg/kg until progression
  * platinum-based chemotherapy (Carboplatin combined with gemcitabine or paclitaxel or pegylated liposomal doxorubicin) will be administrated by intraveinous route at different doses during the induction period x 6 cycles
  Arms: Arm A: Placebo + Avastin + platinum-based chemotherapy

SUMMARY:
This is a phase III, randomized, double-blinded, comparative, multi-centre study to assess the efficacy of atezolizumab in combination with platinum-based chemotherapy plus bevacizumab administered concurrent to chemotherapy and in maintenance, in patients presenting epithelial ovarian cancer (including patients with primary peritoneal and / or fallopian tube adenocarcinoma) who have platinum-sensitive relapse (platinum-free interval > 6 months).

DETAILED DESCRIPTION:
Approximately 600 patients will be randomized using an Interactive Voice Response System /Interactive web system (IVR/IWR system) in a 1:2 ratio to the treatments as specified below:

A. Arm A: Placebo + bevacizumab & platinum-based chemotherapy.

The placebo arm will include one of 3 following regimens up to investigator choice (chosen prior to randomization)

1. Carboplatin (day1)combined with gemcitabine (day1 & day8) and bevacizumab (day1) + placebo ( day1) x 6 cycles q3weeks followed by maintenance with bevacizumab ( day1) + placebo (day1) q3weeks until disease progression or
2. Carboplatin (d1) combined with paclitaxel (day1) and bevacizumab (day1) + placebo (d1) x 6 cycles every 3weeks followed by maintenance with bevacizumab (day1) + placebo (day1) q3weeks until disease progression or
3. Carboplatin (day1) combined with pegylated liposomal doxorubicin (PLD) (day1) and bevacizumab (day1 & 15) + placebo ( day1& 15) x 6 cycles every 4weeks followed by maintenance with bevacizumab (day1) + placebo (day1) q3weeks until disease progression.

B. Arm B: Atezolizumab + bevacizumab & platinum-based chemotherapy

The atezolizumab arm will include one of 3 following regimens up to investigator choice (chosen prior to randomization)

1. Carboplatin (day1) combined with gemcitabine (day1 & d8) and bevacizumab (day1) + atezolizumab ( day1) x 6 cycles q3weeks followed by maintenance with bevacizumab (day1) + atezolizumab (day1) q3w until disease progression or
2. Carboplatin (day1) combined with paclitaxel (day1) and bevacizumab ( day1) + atezolizumab (1200mg, d1) x 6 cycles every 3wk (day1) q3weeks until disease progression or
3. Carboplatin (day1) combined with pegylated liposomal doxorubicin (PLD) (day1) and bevacizumab (day1 & 15) + atezolizumab (day1& 15) x 6 cycles every 4weeks followed by maintenance with bevacizumab (day1) + atezolizumab ( day1) q3weeks until disease progression.

Before randomization to the study:

* A tumor biopsy should have been obtained and sent to the central laboratory
* PD-L1 status should be determined

ELIGIBILITY:
Inclusion Criteria:

1. Female Patients must be ≥18 years of age.
2. Signed informed consent and ability to comply with treatment and follow-up.
3. Patients with histologically confirmed progressive non-mucinous epithelial ovarian cancer, primary peritoneal adenocarcinoma and / or fallopian-tube adenocarcinoma
4. Patients with PD-L1 status determined for stratification on mandatory de novo biopsy sent to central laboratory as a formalin-fixed, paraffin-embedded (FFPE) sample.

   * Cell pellet from pleural effusion, or ascites or lavage are not acceptable.
   * For core needle biopsy specimens, at least three cores should be obtained. Biopsies must be obtained in a manner that minimizes risks. If the location of the tumor renders tumor biopsy medically unsafe or not feasible, patient eligibility should be discussed with the sponsor.
5. Patients whose disease has relapsed more than 6 months from the last dose of platinum before randomization:

   1. criterion for relapse can be according to RECIST v1.1, CA-125 (GCIG) or clinical symptoms
   2. the interval between last dose of platinum and entry in the study should be free of new anti-cancer treatment, with the exception of a maintenance therapy which is allowed up to 21 days before study entry.
6. Patients with one or 2 prior lines of chemotherapy. The last line of chemotherapy should have included platinum.
7. Availability at the study site of representative FFPE tumor sample from surgery during front line therapy, at best before chemotherapy
8. Patients must have normal organ and bone marrow function :

   1. Haemoglobin ≥ 10.0 g/dL.
   2. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L.
   3. Platelet count ≥ 100 x 109/L.
   4. Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN).
   5. Aspartate aminotransferase /Serum Glutamic Oxaloacetic Transaminase (ASAT/SGOT)) and Alanine aminotransferase /Serum Glutamic Pyruvate Transaminase (ALAT/SGPT)) ≤ 2.5 x ULN, unless liver metastases are present in which case they must be ≤ 5 x ULN.
   6. Serum creatinine ≤ 1.5 x institutional ULN,
   7. Patients not receiving anticoagulant medication who have an International Normalized Ratio (INR) ≤1.5 and an Activated ProThrombin Time (aPTT) ≤1.5 x ULN. The use of full-dose oral or parenteral anticoagulants is permitted as long as the INR or APTT is within therapeutic limits (according to site medical standard) and if the patient is on a stable dose of anticoagulants for at least two weeks at the time of randomization.
   8. Urine dipstick for proteinuria < 2+. If urine dipstick is ≥2+, 24-hours urine must demonstrate ≤1 g of protein in 24 hours.
   9. Normal blood pressure or adequately treated and controlled hypertension (systolic BP ≤ 140 mmHg and/or diastolic BP ≤ 90 mmHg).
9. Eastern Cooperative Oncology Group (ECOG) performance status 0-1

For France only: In France, a subject will be eligible for randomization in this study only if either affiliated to, or a beneficiary of, a social security category

Exclusion Criteria:

1. Non-epithelial tumor origin of the ovary, the fallopian tube or the peritoneum (i.e. germ cell tumors).
2. Ovarian tumors of low malignant potential (e.g. borderline tumors)
3. Patients with synchronous primary endometrial cancer unless both of the following criteria are met:

   1. stage < II,
   2. Less than 60 years old at the time of diagnosis of endometrial cancer with stage IA or IB grade 1 or 2, or stage IA grade 3 endometrioid adenocarcinoma OR ≥ 60 years old at the time of diagnosis of endometrial cancer with stage IA grade 1or 2 endometrioid adenocarcinoma.
   3. Patients with serous or clear cell adenocarcinoma or carcinosarcoma of the endometrium are not eligible.
4. Other malignancy within the last 5 years except cervix or breast in situ carcinoma, breast cancer ≥ 3 years free of disease and treatment, type I stage I endometrial cancer).
5. Patients receiving radiotherapy within 6 weeks prior to study treatment.
6. Major surgery within 4 weeks of starting study treatment or patients who have not completely recovered from the effects of any major surgery. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1, Cycle 1
7. Previous allogeneic bone marrow transplant or previous solid organ transplantation.
8. Administration of other simultaneous chemotherapy drugs, any other anticancer therapy or anti-neoplastic hormonal therapy, or simultaneous radiotherapy during the trial treatment period (hormonal replacement therapy is permitted).
9. Prior treatment with CD137 agonists or immune checkpoint blockade therapies, anti-PD1, or anti-PDL1 therapeutic antibodies or anti-CTLA 4.
10. Treatment with systemic immunostimulatory agents (including but not limited to interferon-alpha (IFN-α) and interleukin-2 (IL-2) within 4 weeks or five half-lives of the drug (whichever is shorter) prior to Cycle 1, Day 1
11. Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [TNF] agents) within 2 weeks prior to Cycle 1, Day 1, or anticipated requirement for systemic immunosuppressive medications during the trial

    1. The use of inhaled corticosteroids for chronic obstructive pulmonary disease, mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension, and low-dose supplemental corticosteroids for adrenocortical insufficiency are allowed.
    2. Prophylactic anti-emetic corticosteroids will be avoided if possible in patients treated with pegylated liposomal doxorubicin-carboplatin or gemcitabine-carboplatin regimen. The use of corticosteroids is allowed as premedication for paclitaxel-based regimen and/or premedication in case of carboplatin hypersensitivity.
12. History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with anti-phospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. Are eligible patients with:

    1. a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone
    2. controlled Type 1 diabetes mellitus on a stable insulin regimen
13. History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis. Radiation pneumonitis in the radiation field (fibrosis) detected on screening chest CT scan is permitted
14. Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV). Patients with active hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C.

    Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
15. Signs or symptoms of infection within 2 weeks prior to Cycle 1, Day 1
16. Administration of a live, attenuated vaccine within 4 weeks prior to Cycle 1, Day 1 or anticipation that such a live attenuated vaccine will be required during the study. Influenza vaccination should be given during influenza season only (example approximately October to March in the Northern Hemisphere). Patients must not receive live, attenuated influenza
17. Current or recent (within 10 days prior to randomization) chronic use of aspirin > 325 mg/day.
18. Prior history of hypertensive crisis (CTC-AE grade 4) or hypertensive encephalopathy.
19. Inadequately controlled HTN (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg on antihypertensive medications)
20. Clinically significant (e.g. active) cardiovascular disease, including:

    1. Myocardial infarction or unstable angina within ≤ 6 months of randomization,
    2. New York Heart Association (NYHA) ≥ grade 2 congestive heart failure (CHF),
    3. Poorly controlled cardiac arrhythmia despite medication (patients with rate controlled atrial fibrillation are eligible),
    4. Peripheral vascular disease grade ≥ 3 (e.g. symptomatic and interfering with activities of daily living [ADL] requiring repair or revision)
21. Resting ECG with QTc > 470 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome.
22. Left ventricular ejection fraction defined by MUGA/ECHO below the institutional lower limit of normal (only applicable for patients intended to be treated with pegylated liposomal doxorubicin).
23. Previous Cerebro-Vascular Accident (CVA), Transient Ischemic Attack (TIA) or Sub-Arachnoids Hemorrhage (SAH) within 6 months prior to randomization.
24. History or evidence of hemorrhagic disorders within 6 months prior to randomization.
25. Evidence of bleeding diathesis or significant coagulopathy (in the absence of coagulation).
26. History or clinical suspicion of brain metastases or spinal cord compression. CT/MRI of the brain is mandatory (within 4 weeks prior to randomization) in case of suspected brain metastases. Spinal MRI is mandatory (within 4 weeks prior to randomization) in case of suspected spinal cord compression.
27. History or evidence upon neurological examination of central nervous system (CNS) disease, unless adequately treated with standard medical therapy (e.g. uncontrolled seizures).
28. Significant traumatic injury during 4 weeks prior to randomization.
29. Non-healing wound, active ulcer or bone fracture. Patients with granulating incisions healing by secondary intention with no evidence of facial dehiscence or infection are eligible but require 3 weekly wound examinations.
30. History of VEGF therapy related abdominal fistula or gastrointestinal perforation.
31. Current, clinically relevant bowel obstruction, including sub-occlusive disease, related to underlying disease.
32. Patients with evidence of abdominal free air not explained by paracentesis or recent surgical procedure.
33. Evidence of any other disease, metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment related complications.
34. Women of childbearing potential (<2 years after last menstruation and not surgically sterile) not willing to use highly-effective means of contraception (Appendix 1) during the study and for 6 months after the last dose of study medication
35. Pregnant or lactating women.
36. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
37. Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or to any component of the atezolizumab formulation.
38. Known hypersensitivity reaction or allergy to drugs chemically related to bevacizumab, carboplatin, gemcitabine, paclitaxel, pegylated liposomal doxorubicin, or their excipients that contraindicates the subject's participation

Ages: 18 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 614 (Actual)
Dates: Start 2016-09-22 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
Efficacy: Progression free survival, where the date of progression is based on investigator assessment using the RECIST version 1.1 | An average of 19 months

SECONDARY OUTCOMES:
Efficacy: Overall survival (OS) | To be assessed around 73 months
Efficacy: Time from date randomization to second subsequent therapy or date of death (TSST) whichever come first | To be assessed around 73 months
patient reported outcome variables | to be assessed 19 months
  questionnaire to be completed by patients and collected frequently during the study
Adverse events | to be assessed 19 months
  frequency of adverse events according to MedRA terms

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Emmanuel KURTZ, Principal Investigator — GINECO - Institut de cancérologie Strasbourg Europe
Locations (75):
- Austria (4):
  - Krankenhaus der Barmherzigen Brüder Graz, Graz
  - Medical University of Graz, Graz
  - Medical University of Innsbruck, Innsbruck
  - Medical University of Vienna, Vienna
- Belgium (2):
  - UZ Gent, Ghent
  - Uz Leuven, Leuven
- General University Hospital in Prague, Prague, Czechia
- France (39):
  - ICO Paul Papin, Angers
  - Sainte-Catherine Institut du Cancer Avignon-Provence, Avignon
  - CHRU Jean Minjoz, Besançon
  - Clinique Tivoli, Bordeaux
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Groupe Hospitalier Mutualiste de Grenoble, Grenoble
  - Hôpital Michallon - Centre Hospitalier Universitaire de Grenoble, Grenoble
  - Centre Hospitalier Départemental Les Oudairies, La Roche-sur-Yon
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Hôpital de Mont-de-Marsan, Mont-de-Marsan
  - ICM Val d'Aurelle, Montpellier
  - Centre Azuréen de Cancérologie, Mougins
  - ORACLE - Centre d'Oncologie de Gentilly, Nancy
  - Hôpital Privé du Confluent, S.A.S., Nantes
  - Centre Antoine Lacassagne, Nice
  - CHU Nîmes - Institut de Cancérologie du Gard, Nîmes
  - Centre Hospitalier Régional d'Orléans, Orléans
  - Groupe Hospitalier Diaconesses-Croix Saint Simon, Paris
  - Groupe Hospitalier Saint-Joseph, Paris
  - Hôpital Cochin, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Tenon, Paris
  - Institut Curie - Hopital Claudius Régaud, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre CARIO - HPCA, Plérin
  - Hôpital de la Milétrie - Centre Hospitalier Universitaire de Poitiers - Pôle Régional de Cancérologie, Poitiers
  - Centre Eugène Marquis, Rennes
  - Hôpital René Huguenin, Institut Curie, Saint-Cloud
  - ICO Centre René Gauducheau, Saint-Herblain
  - Centre Paul Strauss, Strasbourg
  - Institut de Cancérologie Strasbourg Europe (ICANS), Strasbourg
  - Clinique Pasteur, Toulouse
  - Institut Claudius Regaud, Toulouse
  - ICL Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif
- Germany (16):
  - Charité, Campus Virchow-Klinikum, Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Universitatsklinikum Dusseldorf, Düsseldorf
  - Kliniken Essen Mitte, Evang. Huyssens-Stiftung, Essen
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Jena, Jena
  - Städtisches Klinikum Karlsruhe, Karlsruhe
  - Klinikum der Universität München - LMU, Campus Großhadern, München
  - Klinikum rechts der Isar, Technischen Universität München, München
  - Sana Klinikum Offenbach, Offenbach
  - Studienzentrum Onkologie Ravensburg, Ravensburg
  - Universitatsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - Klinikum Worms, Worms
- Sharre Zedek Medical Centre, Jerusalem, Israel
- Spain (12):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínic Barcelona, Barcelona
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital Universitari de Girona ICO Girona (Dr. Josep Trueta), Girona
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Central Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario Son Espases, Palma de Mallorca
  - Hospital Universitario Donostia, San Sebastián
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Alvaro Cunqueiro, Vigo

REFERENCES:
- [Derived] Kurtz JE, Pujade-Lauraine E, Oaknin A, Belin L, Leitner K, Cibula D, Denys H, Rosengarten O, Rodrigues M, de Gregorio N, Martinez Garcia J, Petru E, Kocian R, Vergote I, Pautier P, Schmalfeldt B, Gaba L, Polterauer S, Mouret Reynier MA, Sehouli J, Churruca C, Selle F, Joly F, D'Hondt V, Bultot-Boissier E, Lebreton C, Lotz JP, Largillier R, Heudel PE, Heitz F; ATALANTE/ENGOT-ov29 Investigators. Atezolizumab Combined With Bevacizumab and Platinum-Based Therapy for Platinum-Sensitive Ovarian Cancer: Placebo-Controlled Randomized Phase III ATALANTE/ENGOT-ov29 Trial. J Clin Oncol. 2023 Oct 20;41(30):4768-4778. doi: 10.1200/JCO.23.00529. Epub 2023 Aug 29. PMID 37643382